CLINICAL TRIAL: NCT00559377
Title: A Phase 2 Study of Positron Emission Tomography Imaging With [18F]-Fluoromisonidazole (FMISO) and [18F]-Fluorodeoxyglucose (FDG) for Assessment of Tumor Hypoxia in Cervical Cancer
Brief Title: FDG and FMISO PET Hypoxia Evaluation in Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCI-2009-00257; NCI-2009-00257 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UW IRB# 6143 (Other: University of Washington Medical Center); 7958 (Other: CTEP); N01CM37008 (NIH)
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Results first posted 2015-06-26 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Cervical Adenocarcinoma; Cervical Squamous Cell Carcinoma; Stage IB Cervical Cancer; Stage IIA Cervical Cancer; Stage IIB Cervical Cancer; Stage III Cervical Cancer; Stage IVA Cervical Cancer; Stage IVB Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — fluoromisonidazole; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic FMISO AND FDG PET (Experimental): Patients receive ^18F FMISO IV over 1 minute followed by PET scanning. Patients undergo a second ^18F FMISO PET scan 4-8 weeks later. Patients who have not had a prior ^18F FDG PET scan as part of their routine clinical management undergo ^18F FDG PET scanning at baseline.
  Interventions: Other: 18F-fluoromisonidazole; Radiation: fluorodeoxyglucose F 18; Procedure: positron emission tomography; Other: tissue oxygen measurement

INTERVENTIONS:
Other: 18F-fluoromisonidazole — Undergo ^18F FMISO PET scan
  Other Names: 18F-FMISO
Radiation: fluorodeoxyglucose F 18 — Undergo ^18F FDG PET scan
  Other Names: 18FDG; FDG
Procedure: positron emission tomography — Undergo ^18F-FMISO and ^18F FDG PET scan
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Other: tissue oxygen measurement — Undergo ^18 F FMISO PET and ^18F FDG PET

SUMMARY:
This phase II trial is studying how well PET scans using fluoromisonidazole F 18 and fludeoxyglucose F 18 work in finding oxygen in tumor cells of patients undergoing treatment for newly diagnosed stage 1B, stage II, stage II, or stage IV cervical cancer. Diagnostic procedures using positron emission tomography (PET scan), fluoromisonidazole F 18, and fludeoxyglucose F 18 to find oxygen in tumor cells may help doctors predict how patients will respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Test the extent to which fluoromisonidazole F 18 ([^18F] FMISO) uptake predicts survival of patients undergoing therapy for newly diagnosed stage IB-IVB cervical cancer.

SECONDARY OBJECTIVES:

I. Test [^18F] FMISO tumor uptake as an independent predictor of response to therapy and that it provides additional predictive power over fludeoxyglucose F 18 ([^18F] FDG).

II. Test [^18F] FMISO tumor uptake as a predictor of response in a subgroup of patients receiving radiotherapy.

III. Test the relationship between [^18F] FMISO uptake in the primary tumor and the volume of the primary tumor estimated by CT scan.

IV. Test the reproducibility of [^18F] FMISO uptake in tumors by imaging the same patients on sequential days in a test-retest protocol.

V. Compare [^18F] FMISO PET or PET/CT scan with [^18F] FDG PET or PET/CT scan to test whether [^18F] FMISO is an independent predictor of treatment outcome.

OUTLINE:

Patients receive fluoromisonidazole F 18 ([^18F] FMISO) IV over 1 minute followed by PET scanning. Patients undergo a second [^18F] FMISO PET scan 4-8 weeks later. Patients who have not had a prior fludeoxyglucose F 18 ([^18F] FDG) PET scan as part of their routine clinical management undergo [^18F] FDG PET scanning at baseline. A subset of 10 patients undergo two [^18F] FMISO PET scans within a 48-hour period to evaluate the variability (test-retest) of this imaging measurement.

Patients response to therapy is followed periodically until time to disease progression or for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell or adenocarcinoma of the uterine cervix
* Clinical stage IB-IVB by FIGO criteria

  * Size of the primary tumor ≥ 2 cm as assessed by CT scan
* Measurable disease
* Scheduled to undergo radiotherapy, chemotherapy, or combined multimodality management
* No prior cervical cancer diagnosis
* No known brain metastases
* ECOG performance status (PS) 0-2 (Karnofsky PS 60-100%)
* Life expectancy > 12 months
* Not pregnant
* No nursing for 24 hours after fluoromisonidazole F 18 ([^18F] FMISO) PET scanning
* Negative pregnancy test
* Weight ≤ 400 lbs
* Sufficiently healthy to undergo cancer treatment
* Willing to undergo PET scanning with urinary bladder catheterization
* Leukocytes ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin normal
* AST/ALT ≤ 2.5 times normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* No serious medical co-morbidities that would preclude definitive local therapy
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to [^18F] FMISO
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements.
* No prior surgery or radiotherapy for cervical cancer
* Other concurrent investigational agents allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-11; Primary Completion 2012-07 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Rajendran, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic (^18F FMISO PET and ^18F FDG PET): Patients receive ^18F FMISO IV followed by PET scanning. Patients undergo a second ^18F FMISO PET scan 4-8 weeks later. Patients who have not had a prior ^18F FDG PET scan as part of their routine clinical management undergo ^18F FDG PET scanning at baseline.
Period: Overall Study
Arm/Group | Diagnostic (^18F FMISO PET and ^18F FDG PET)
Started | 16
Completed | 7
Not Completed | 9
Not completed — Withdrawal by Subject | 9

BASELINE CHARACTERISTICS:
Groups:
- All Patients: Patients receive ^18F FMISO IV followed by PET scanning. Patients undergo a second ^18F FMISO PET scan 4-8 weeks later.
Arm/Group | All Patients
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Evaluate the value of pre-treatment FMISO results (T:B and HV) for all patients to predict the survival outcome variables.
Time Frame: For up to 2 years
Population: 1 patient has been lost to follow up for survival measures.
Measure: Number; unit: participants still alive after 2 years
Groups:
- 2 Year Overall Survival: Patients who have not been declared deceased for 2 years after their last FMISO scan.
Arm/Group | 2 Year Overall Survival
Number analyzed (Participants) | 15
participants still alive after 2 years | 11
Statistical Analysis 1: Comparison: 2 Year Overall Survival; This outcome is for comparing FMISO Hypoxic Volume to overall survival; Test type: Superiority or Other; p = .42, Regression, Cox; Hazard Ratio (HR) = 1.27
Statistical Analysis 2: Comparison: 2 Year Overall Survival; This outcome is for comparing FMISO T:Bmax to overall survival; Test type: Superiority or Other; p = .87, Regression, Cox; Hazard Ratio (HR) = 1.05

2. Primary Outcome: Disease-free Survival (DFS)
Description: Evaluate the value of pre-treatment FMISO results (T:B and HV) for all patients to predict the disease free survival outcome variables.
Time Frame: Up to 2 years
Population: Of the 13 patients analyzed for disease-free survival, 10 remained disease-free throughout the 2 year follow up. For 3 patients, we could determine overall survival, but could not confirm whether or not they were disease-free.
Measure: Number; unit: participants disease-free after 2 years
Groups:
- Disease-Free Survival: Patients who have remained disease-free throughout the 2 year follow up
Arm/Group | Disease-Free Survival
Number analyzed (Participants) | 13
participants disease-free after 2 years | 10
Statistical Analysis 1: Comparison: Disease-Free Survival; This outcome is for comparison of FMISO Hypoxic Volume to disease-free survival; Test type: Superiority or Other; p = .58, Regression, Cox; Hazard Ratio (HR) = 1.18
Statistical Analysis 2: Comparison: Disease-Free Survival; This outcome is for comarison of FMISO T:Bmax to progression-free survival; Test type: Superiority or Other; p = .98, Regression, Cox; Hazard Ratio (HR) = .99

3. Secondary Outcome: Relationship Between Hypoxia-related IHC Biomarkers and Regional FMISO Uptake in Tumor
Description: The value of the biomarker by IHC analyses relates primarily to validating the information content of FMISO images.
Time Frame: Up to 2 years
Population: 11 tissue samples with Hif1, VEGF, p53 and EGFR IHC values were compared to FMISO uptake.
Measure: Median (Full Range); unit: units on a scale 0=low, 8=high
Groups:
- Patients With IHC Measures: Patients who had tissue used to evaluate immunohistochemistry measures correlated to FMISO uptake where IHC scores were calculated by standard Allred values.
Arm/Group | Patients With IHC Measures
Number analyzed (Participants) | 11
units on a scale 0=low, 8=high
  Hif1 | 5 [3 to 7]
  VEGF | 5 [0 to 7]
  p53 | 7 [4 to 8]
  EGFR | 7 [3 to 8]
Statistical Analysis 1: Comparison: Patients With IHC Measures; The correlation between IHC values and FMISO uptake were analyzed using Spearman correlation where p values less than 0.05 were considered significant; Test type: Superiority or Other; p < 0.05, Spearman Correlation; Spearman Correlation = .004

4. Secondary Outcome: Relationship Between Ki67 and Regional FMISO Uptake in Tumor
Description: The value of the biomarker Ki67 analyses relates primarily to validating the information content of FMISO images.
Time Frame: Up to 2 years
Population: 11 tissue samples with Ki67 values were compared to FMISO uptake.
Measure: Mean (Standard Deviation); unit: percentage of staining
Arm/Group | Patients With IHC Measures
Number analyzed (Participants) | 11
percentage of staining | 74 (18)

5. Secondary Outcome: Response to XRT Using RECIST
Description: Response for the XRT is evaluated by the radiation oncologists as per standard clinical protocols
Time Frame: time to disease progression or 2 years following first FMISO scan
Population: PET/CT acquisition was obtained using non-diagnostic low dose CT attenuation scans at the time of PET/CT imaging that limited our ability to accurately measure tumor dimensions and due to lack of complete data, we were not able to fulfill this aim.
Arm/Group | Patients Who Had Response Determined by Clinical RECIST
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: As a PET imaging study, AEs are assessed at 3 hours post injection (end of the scan) and up to 10 hours following the scan
Arm/Group | Diagnostic (^18F FMISO PET and ^18F FDG PET)
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

LIMITATIONS AND CAVEATS:
Small number of subjects enrolled and events limit meaningful statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less